CLINICAL TRIAL: NCT01230216
Title: Effect of Intensive Blood Pressure Control on Progression of Coronary Atherosclerosis: Randomized Evaluation by Intravascular Ultrasound
Acronym: PREVUS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow patients enrollment
Sponsor: Takeshi Morimoto (Other)
Responsible Party: Sponsor-Investigator, Takeshi Morimoto, Professor, Kyoto University, Graduate School of Medicine
Organization: Kyoto University, Graduate School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C464
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Disease; Hypertension
Keywords: coronary artery disease; hypertension
MeSH Terms: conditions — Coronary Artery Disease; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intensive blood pressure control (Active Comparator): systolic blood pressure less than 120 mmHg
  Interventions: Drug: control systolic blood pressure less than 120 mmHg
- standard blood pressure control (Active Comparator): systolic blood pressure less than 140 mmHg
  Interventions: Drug: control systolic blood pressure less than 140 mmHg

INTERVENTIONS:
Drug: control systolic blood pressure less than 120 mmHg — use losartan to control blood pressure
  Arms: intensive blood pressure control
Drug: control systolic blood pressure less than 140 mmHg — use losartan to control blood pressure
  Arms: standard blood pressure control

SUMMARY:
The purpose of this study is to evaluate the effect of intensive blood pressure control compared to standard blood pressure control on progression of coronary atherosclerosis by intravascular ultrasound in hypertensive patients with coronary artery disease.

DETAILED DESCRIPTION:
Antihypertensive therapy is reported to reduce cardiovascular events in patients with coronary artery disease. The goal of blood pressure in patients with coronary artery disease is recommended to control below 140/90mmHg. However, the effect of intensive blood pressure control compared to standard blood pressure control is still unknown. The purpose of this study is to evaluate the effect of intensive blood pressure control compared to standard blood pressure control on progression of coronary atherosclerosis by intravascular ultrasound in hypertensive patients with coronary atherosclerosis after 18 months. The goal of systolic blood pressure is under 120mmHg in intensive blood pressure control group and under 140mmHg in standard blood pressure control group. The design of this study is randomized control study.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery diseases which require coronary angiography or percutaneous coronary intervention
* primary hypertension (systolic blood pressure 140-180mmHg within one month)

Exclusion Criteria:

* severe hypertension
* secondary hypertension
* treated with more than three antihypertensive drugs
* left main trunk trunk coronary artery disease
* moderate heart failure
* severe valvular disease
* liver dysfunction renal dysfunction (Cr>=2.0mg/dl) Pregnant or nursing women severe arrhythmia

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-12; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
change of percent atheroma volume | 1.5-year
  change of percent atheroma volume measured by intravascular ultrasound

SECONDARY OUTCOMES:
all cause death | 1.5-year
  Death from any cause
cardiac death | 1.5-year
  Death from cardiac diseases
cardiovascular death | 1.5-year
  Death from cardiovascular diseases
myocardial infarction | 1.5-year
  myocardial infarction defined by ARC
stroke | 1.5-year
  both ischemic and hemorrhagic strokes excluding transient ischemic attack
target-lesion revascularization | 1.5-year
  target-lesion revascularization
any coronary revascularization | 1.5-year
  any coronary revascularization
hospitalization due to angina pectoris | 1.5-year
  hospitalization due to angina pectoris
hospitalization due to heart failure | 1.5-year
  hospitalization due to heart failure
change of total atheroma volume | 1.5-year
  change of total atheroma volume measured by intravascular ultrasond
percent change of total atheroma volume | 1.5-year
  percent change of total atheroma volume measured by intravascular ultrasound
change of atheroma volume at most severe 10mm lesion | 1.5-year
  change of atheroma volume at most severe 10mm lesion measured by intravascular ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, PhD, Principal Investigator — Professor of Medicine, Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Division of Cardiology, Kyoto University Hospital, Kyoto, Kyoto, Japan

REFERENCES:
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623